CLINICAL TRIAL: NCT03255694
Title: A Phase 2 Study Extension Period of Pegylated Somatropin (PEG-somatropin) in the Treatment of Children With Idiopathic Short Stature: An Open, Non-controlled Observational Study.
Brief Title: A Study Extension Period of PEG-somatropin (Pegylated-somatropin) in the Treatment of Children With Idiopathic Short Stature
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other); The First Hospital of Jilin University (Other); Affiliated Hospital of Jiangnan University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanghai Children's Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Children's Hospital of Fudan University (Other); Jiangxi Province Children's Hospital (Other); Hunan Children's Hospital (Other Government); Beijing Children's Hospital (Other); Children's Hospital of Soochow University (Other); Wuxi Women's & Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 033 CT-Extension Period
Record Dates: First submitted 2017-07-14; First posted 2017-08-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Dwarfism
MeSH Terms: conditions — Dwarfism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEG-somatropin (Experimental): After the first stage (52 weeks) of Phase II clinical trial, the initial medication dose of this extension period is 0.2 mg/kg weight/week of PEG-rhGH for the high dose group, low dose group and negative control group, and it is adjusted in accordance with yearly height velocity (HV) and IGF-1 SDS of each visit. The maximum dose shall not exceed 0.4 mg/kg weight/week.
  Interventions: Drug: PEG-somatropin

INTERVENTIONS:
Drug: PEG-somatropin — After the first stage (52 weeks) of Phase II clinical trial, the initial medication dose of this extension period is 0.2 mg/kg weight/week of PEG-rhGH for high dose group, low dose group and negative control group, and it is adjusted in accordance with yearly height velocity (HV) and IGF-1 SDS of each visit. The maximum dose shall not exceed 0.4 mg/kg weight/week.
  Other Names: Polyethylene Glycol Recombinant Human Somatropin Injection

SUMMARY:
After the first stage (52 weeks) of Phase II clinical trial, Pegylated recombinant human growth hormone (PEG-rhGH) injection of appropriate dose in compliance with ISS clinical treatment strategy is used to treat children with ISS (Idiopathic Short Stature). The long-term efficacy and safety of the investigational product are evaluated, which can provide more scientific and reliable medication guidance information for clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who have completed the first stage (52 weeks) of Phase II clinical trial (including negative controls) with completed follow-up records may be enrolled in the extension period study.
* Before the extension period study, the investigator shall fully inform the subjects and their guardians of all the information about the extension period study, including detailed follow-up procedure, treatment plan, laboratory examination items during follow-ups and possible benefits and risks. The extension period study shall only be initiated after the subjects and their guardians are well informed, and agree to cooperate and complete the treatment, follow-ups and examinations during the study, and sign the written informed consent.

Exclusion Criteria:

* Subjects who have taken the following medications within 2 months before entering the extension period study:

  1. Aromatase inhibitors (which include but are not limited to Lelrozol and Anastrozole), with continuous medication ≥1 month;
  2. Gonadotropin releasing hormone analogues (which include but are not limited to Triptorelin, Leuprorelin and Goserelin),, with continuous medication ≥1 month;
  3. Sex steroids (which include but are not limited to any type of estrogen, progestin and androgen) , with continuous medication ≥1 month;
  4. Protein anabolic drugs (which include but are not limited to Oxandrolone, Danazol and Strombafort), with continuous medication ≥1 month;
  5. Glucocorticoids via oral/intravenous administration for more than 1 month..

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change of yearly height velocity (ΔHV) | Baseline，the end of 3-year addendum
  Change of yearly height velocity before and after treatment. Yearly Height Velocity=12×(Height Yx - Height at Baseline)/(Date of Yx - Date of Baseline)(Yx refers to the height value at particular timepoint x)

SECONDARY OUTCOMES:
Standard deviation score of height at the actual age (ΔHT SDS) | Baseline，every 3 months，the end of 3-year addendum
  Standard deviation score of height at the actual age.
Change fo Bone maturation | Baseline，every 3 months，the end of 3-year addendum
  Change fo Bone maturation before and after treatement (bone age/chronological age)
Change of IGF-1 SDS (ΔIGF-1 SDS) | Baseline，every 3 months，the end of 3-year addendum
  Change of IGF-1 SDS before and after treatement
Changes of standard deviation scores of body mass index (ΔBMI SDS) | Baseline，every 3 months，the end of 3-year addendum
  Changes of standard deviation scores of body mass index
The yearly average dose of PEG-rhGH injection | Baseline，every 3 months，the end of 3-year addendum
Final height (FH) | Baseline，every 3 months，the end of 3-year addendum
  Final height
The improvement of FH compared with the baseline predicted adult height (PAH) | Baseline，every 3 months，the end of 3-year addendum
Improvement of NAH (near adult height) | Baseline，every 3 months，the end of 3-year addendum
  For subjects who reach NAH with treatment but fail to follow-ups before reaching FH, the improvement of NAH in comparison with the baseline PAH (predicted adult height) shall be evaluated
the improvement of PAH | Baseline，every 3 months，the end of 3-year addendum
  For subjects who fail to reach NAH with treatment and fail to follow-ups before reaching FH, the improvement of PAH in comparison with the baseline PAH shall be evaluated
The changes of the scores evaluated by the Quality of Life Scale | Baseline，every 3 months，the end of 3-year addendum
The changes of lean body mass (LBM) (optional) | Baseline，every 3 months，the end of 3-year addendum
The changes of fat mass (torso) (FM) (optional) | Baseline，every 3 months，the end of 3-year addendum
The changes of the percentage of body fat (optional) | Baseline，every 3 months，the end of 3-year addendum
The changes of bone mineral density (BMD) (optional) | Baseline，every 3 months，the end of 3-year addendum

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, Principal Investigator — Department of Pediatrics of Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (12):
- China (12):
  - Beijing Children's Hospital, Capital Medical University, National Center for Children's Health, Beijing, Beijing Municipality
  - Department of Pediatrics of Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Children's Hospital of Soochow University, Naning, Jiangsu
  - The First Affiated Hospital of Nanjing Medical Universit, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Wuxi Children's Hospital, Wuxi, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Shanghai Children's Hospital of Fudan University, Shanghai
  - Shanghai Children's Hospital, Shanghai